CLINICAL TRIAL: NCT02422719
Title: Radotinib Efficacy and Safety Validation in Chronic Phase Chronic Myeloid Leukemia Patients Who Are Intolerant or Resistant to at Least Two Tyrosine Kinase Inhibitors As a Third or Subsequent Line Therapy
Brief Title: Radotinib as 3rd or Later Line Therapy in CP-CML
Acronym: REVITAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Hawk Kim, Associate Professor, Ulsan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD-201501
Record Dates: First submitted 2015-04-05; First posted 2015-04-21 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; Intolerance; Resitance; Radotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — 4-methyl-N-(3-(4-methylimidazol-1-yl)-5-trifluoromethylphenyl)-3-(4-pyrazin-2-ylpyrimidin-2-ylamino)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radotinib (Experimental): Radotinib treatement single arm
  Interventions: Drug: Radotinib

INTERVENTIONS:
Drug: Radotinib — Radotinib 400mg bid
  Other Names: Supect

SUMMARY:
The purpose of this study is to determine whether radotinib is effective and safe for patients with chronic myeloid leukemia, chronic phase who are intolerable or resistant to prior 2 or more tyrosine kinase inhibitors.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether radotinib 400mg bid is effective and safe for patients with chronic myeloid leukemia, chronic phase who are intolerable or resistant to prior 2 or more tyrosine kinase inhibitors. The primary end point is major cytogenetic response by 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronic myeloid leukemia chronic phase (CP-CML) patients who are not tolerable or resistant to prior 2 or more tyrosine kinase inhibitors (TKIs).
* ECOG 0, 1, 2
* Patients who are agree and signed to informed consent.

Exclusion Criteria:

* T315I mutation
* Prior exposure to radotinib
* Accelerated or blastic phase
* galactose intolerance, severe lactase deficiency or glucose galactose malabsorption
* Prior history of intensive cytotoxic chemotherapy except for TKIs
* Significant cardiac problem
* QTcF > 450 msec
* Pancreatitis history prior to study enrollment
* Clinically significant malignant disease other than CML
* Pregnant or breast feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Major cytogenetic response | by 12 months after radotinib treatment
  The rate of achieving major cytogenetic response [35% or less t(9;22) chromosome by conventional banding technique] in bone marrow by 12 months after radotinib treatment will be the primary end point.

SECONDARY OUTCOMES:
Rate of Major Molecular response (MR3.0) on each time point | up to 12 months
The number of Participants with Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hawk Kim, M.D., Ph.D., Principal Investigator — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea